CLINICAL TRIAL: NCT05836779
Title: A Phase 2a, Open Label Study to Evaluate the Safety, Tolerability, and Efficacy of CBL-514 Injection for the Treatment of Edematous Fibrosclerotic Panniculopathy (EFP) Cellulite (Stage 2)
Brief Title: A Study to Evaluate the Efficacy and Safety of CBL-514 in Participants With EFP; Cellulite (Stage 2)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Caliway Biopharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CBL-0201EFP (Stage 2)
Record Dates: First submitted 2023-04-19; First posted 2023-05-01 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Cellulite
MeSH Terms: conditions — Cellulite

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CBL-514 up to 320mg (Experimental): Participants will receive up to 320 mg per treatment session at intervals of approximately 4 weeks for up to a maximum of 2 treatments.
  Interventions: Drug: CBL-514 injection

INTERVENTIONS:
Drug: CBL-514 injection — CBL-514 will be administered at the raised area of cellulite.

SUMMARY:
The Stage 2 of this phase 2 study is an open-label, single-arm study to assess the efficacy and safety of CBL-514 in participants with Edematous Fibrosclerotic Panniculopathy (EFP) cellulite.

DETAILED DESCRIPTION:
This Phase 2a study has an integrated design consisting of a single ascending dose (SAD) part in Stage 1 followed by a single-arm design in Stage 2. The Stage 2 will include a total of 20 participants enrolled in 1 selected CBL-514 dose.

Eligible participants will be sequentially assigned to receive up to 2 courses of allocated CBL-514 dose administered by subcutaneous injection on both sides of the posterolateral thighs.

ELIGIBILITY:
Inclusion Criteria:

1. Female aged 18 years to 64 years old (at Screening), inclusive.
2. Have a BMI > 18.5 and < 35 kg/m2 and body weight ≥ 50 kg at Screening and Day 1.
3. The participant has both sides of posterolateral thighs assessed according to the modified Hexsel CSS (A) number of evident depressions, (B) depression depth scale, and (C) morphological appearance of skin surface alterations. On assessment by the modified Hexsel CSS, the participant scores at least 4 and no greater than 8 at Screening and Day 1.

   The total score must contain:
   1. Hexsel CSS item (A) 'number of evident depressions' score of ≥1
   2. Hexsel CSS item (B) 'depth of depressions' score of ≥ 1
4. Participant has a stable lifestyle (e.g., exercise, eating patterns, and smoking habit) per participant report for at least 3 months before Screening and during the study.
5. Voluntarily signs the informed consent form and, in the opinion of the Investigator or delegate, is physically and mentally capable of participating in the study, and willing to adhere to study procedures.

Exclusion Criteria:

1. Female participant of childbearing potential who is not willing to commit to an acceptable contraceptive regimen with her partner from the time of Screening and throughout study participation until 90 days after the last IP dose, or who is currently pregnant or lactating. Note: females who are not of childbearing potential are not required to use contraception. Females not of childbearing potential are defined as those who have been surgically sterilized (hysterectomy or bilateral oophorectomy) or who are postmenopausal (defined as aged at least 50 years old with ≥ 12 months of amenorrhea and a follicle-stimulating hormone [FSH] > 30 IU/L at Screening).
2. Participant diagnosed with coagulation disorders or is receiving anticoagulant/antiplatelet therapy or medications or dietary supplements, which impede coagulation or platelet aggregation within 14 days prior to the IP administration.
3. Participant has hemoglobin A1c (HbA1c) ≥ 9%, delayed wound healing, or any diabetic risks which, in the opinion of the Investigator (or designee) is inappropriate to participate in the study.
4. Participant has a clinically significant cardiovascular disease and abnormal findings in electrocardiogram (ECG) at Investigator's (or designee's) discretion.
5. Participant with active or prior history of malignancies within 5 years before Screening or being assessed for a possible malignancy. Except adequately treated basal cell carcinoma of the skin and in situ squamous cell carcinoma of the skin would be eligible as per Investigator's (or designee's) discretion.
6. Participant with a history of human immunodeficiency virus (HIV)-1 infection, or participants with active HIV infection at Screening with a positive HIV antigen/antibody (Ag/Ab) combination test.
7. Participant with a history of trypanophobia, the extreme fear of medical procedures involving injections or needles, or who experience vasovagal syncope and pass out at the sight of blood or a needle.
8. Participant with any hepatic medical condition that, in the opinion of the Investigator (or designee), would interfere with assessment of safety or efficacy or compromise the participant's ability to undergo study procedures or provide informed consent.
9. Participant who has a recent history of major depression, anxiety, or other psychiatric disease requiring treatment with prescription medication within 6 months prior to Screening.
10. Participant has abnormal skin or local skin conditions at the treatment area, which in the opinion of the Investigator (or designee), is inappropriate to participate in the study. This includes but is not limited to any of the following:

    1. skin manifestations of a systemic disease
    2. any abnormality of the skin or soft tissues on the anticipated treatment area
    3. skin laxity on treatment area when the participant is in the standing position
    4. sensory loss or dysesthesia in the area to be treated
    5. evidence of any cause of enlargement in the area to be treated other than localized subcutaneous fat
    6. tattoos on the area to be treated
    7. participant with a propensity for keloid or hypertrophic scarring.
11. Participant who has had the following surgical or aesthetic procedures:

    1. liposuction, cryolipolysis, ultrasonic lipolysis, low level laser therapy (LLLT), or lipolysis injection to the region to be treated before Screening
    2. medical device, injection (including but not limited to collagenase clostridium histolyticum injections and collagen stimulating injections), over-the-counter (OTC) cosmetic cream, or cosmetic program to prevent or mitigate EFP to the region to be treated within 12 months before Screening and throughout study participation
    3. massage to the region to be treated within 2 weeks before Screening and throughout study participation.
12. Participant is undergoing chronic steroid or immunosuppressive therapy, except for asthma inhaler or topical steroids for skin conditions if the medications are not used on the treatment area.
13. Participating is requiring continual use of the following therapeutic agents during the study: terfenadine, buspirone, fexofenadine, any medication that is known to strongly inhibit or induce CYP enzymes, sensitive CYP substrates or drugs with narrow therapeutic index, which in the opinion of the Investigator (or designee), may affect the evaluation of the investigational product or place the participant at undue risk. If a participant needs to use the above-mentioned therapeutic agents during the study for any reason, these therapeutic agents should not be used at least for 2 days before dosing and until 1 day after dosing.
14. Participant receives nonsteroidal anti-inflammatory drug (NSAID) including aspirin within 14 days prior to the IP administration.
15. Participant is unable to receive topical anesthesia (e.g., history of hypersensitivity to lidocaine).
16. Participant with known allergies or sensitivities to the IP or its components.
17. Participant with liver cirrhosis or with inadequate liver function at Screening defined as aspartate aminotransferase (AST), alanine aminotransferase (ALT), alkaline phosphatase (ALKP), total bilirubin(TBIL), or gamma-glutamyl transferase (GGT) > 3.0 × upper limit of normal (ULN).
18. Participant with any renal impairment, defined as abnormal serum creatinine, and urea > 1.5 × ULN or estimated glomerular filtration rate (eGFR) < 90 mL/min/1.73 m2. Participants who are currently on dialysis should be excluded.

    Participants with an eGFR ≥ 60 and < 90 mL/min/1.73 m2 at Screening should be evaluated by the Investigator to exclude pre-existing renal disease or associated dysfunction. If mild decrease in eGFR is assessed by the Investigator as not clinically significant or not related to dysfunction, the participants may be eligible upon the Investigator's assessment.
19. Use of other investigational product or device within 4 weeks prior to Screening.

Ages: 18 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2023-05-10 (Actual); Primary Completion 2023-11-29 (Actual); Study Completion 2024-01-05 (Actual)

PRIMARY OUTCOMES:
Evaluation of the score change of edematous fibrosclerotic panniculopathy (EFP) measured by cellulite severity scale from baseline following administration of at least 1 course of CBL-514. | 4 weeks from the final treatment visit
  Change in total scores from baseline according to the modified Hexsel CSS at V4 based on (A) number of evident depressions, (B) depression depth scale, and (C) morphological appearance of skin surface alterations following administration of at least 1 course of CBL-514.
  (A) Number of evident depressions: '0' = None/no depressions '1' = 1 to 4 depressions are visible '2' = 5 to 9 depressions are visible '3' = 10 or more depressions are visible (B) Depth of depressions: '0' = No depressions '1' = Superficial depressions '2' = Medium depth depressions '3' = Deep depressions (C) Morphological appearance of skin surface alterations: '0' = No raised areas '1' = 'Orange peel' appearance '2' = 'Cottage cheese' appearance '3' = 'Mattress' appearance
  The total score of (A), (B) and (C) will determine the cellulite severity level as follows :
  0 = None 1-3 = Mild 4-6 = Moderate 7-9 = Severe

SECONDARY OUTCOMES:
Percentage of participants' thighs that achieve at least 1-level severity improvement measured by cellulite severity scale from baseline following administration of 1 course of CBL-514. | Up to 12 weeks from the final treatment visit
  Percentage of participants' thighs with at least 1-level severity improvement determined by the total scores of modified Hexsel CSS at V4 and V5 compared to baseline.
Evaluation of the total score change of edematous fibrosclerotic panniculopathy (EFP) measured by cellulite severity scale from baseline following administration of at least 1 course of CBL-514. | 12 weeks from the final treatment visit
  Change in total scores according to the modified Hexsel CSS at V5.
Percentage of participants' thighs that achieve at least 2-score improvement measured by cellulite severity scale from baseline following administration of 1 course of CBL-514. | Up to 12 weeks from the final treatment visit
  Percentage of participants' thighs with achieve at least 2-score improvement in modified Hexsel CSS at V4 and V5.
Evaluation of the response rate of EFP score change by Global Aesthetic Improvement Scale (GAIS) reported by the clinician and participant, respectively, following the administration of at least 1 course of CBL-514. | Up to 12 weeks from the final treatment visit
  Percentage of participants with a score change in GAIS assessed by the clinician and participant, respectively.

OTHER OUTCOMES:
Incidence of adverse events and treatment-emergent adverse events (TEAEs) | Up to 12 weeks from the final treatment visit
  Number of participants experiencing TEAEs and number of individual TEAEs
Incidence of adverse events and treatment-emergent adverse events (TEAEs) at the injection site(s) | Up to 12 weeks from the final treatment visit
  Number of participants experiencing TEAEs and number of individual TEAEs at the injection site(s)
Incidence of adverse events and treatment-emergent adverse events (TEAEs) related to the investigational product (IP) | Up to 12 weeks from the final treatment visit
  Number of participants experiencing TEAEs and number of individual TEAEs related to the investigational product (IP)
Incidence of adverse events of special interest | Up to 12 weeks from the final treatment visit
  Number of participants experiencing adverse events of special interest
Number of participants with clinically significant abnormalities in laboratory tests | Up to 12 weeks from the final treatment visit
  Laboratory tests include assessment of hematology, biochemistry, coagulation, and urinalysis tests
Number of participants with clinically significant abnormalities in physical examination | Up to 12 weeks from the final treatment visit
  Physical examinations include assessment of 12-lead electrocardiogram parameters and vital signs
Incidence of use of concomitant medications to treat treatment-emergent adverse events (TEAEs) | Up to 12 weeks from the final treatment visit
  Number of participants experiencing use of concomitant medications to treat treatment-emergent adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Anne Sheu, Study Director — Caliway Biopharmaceuticals Co., Ltd.
Locations (5):
- United States (5):
  - Investigational Site 6, Encinitas, California
  - Investigational Site 1, Encino, California
  - Investigational Site 3, San Diego, California
  - Investigational Site 4, Coral Gables, Florida
  - Investigational Site 2, New York, New York